CLINICAL TRIAL: NCT00486876
Title: A Double-Blind, Randomized, Placebo-Controlled Phase 2b Study of 100, 200, and 300 mg BID Dextofisopam in Female Outpatients With Irritable Bowel Syndrome
Brief Title: A Study of 3 Doses of Dextofisopam in Females With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmos (Industry)
Responsible Party: President, Pharmos Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VPI-TOFP-203
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Diarrhea predominant Irritable Bowel Syndrome; Alternating Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — tofisopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Dextofisopam
- 2 (Experimental): 100 mg BID
  Interventions: Drug: Dextofisopam
- 3 (Experimental): 200 mg BID
  Interventions: Drug: Dextofisopam
- 4 (Experimental): 300 mg BID
  Interventions: Drug: Dextofisopam

INTERVENTIONS:
Drug: Dextofisopam — capsules, 0 (placebo), 100, 200, and 300 mg BID for 12 weeks

SUMMARY:
The primary objectives of this study are to evaluate the clinical safety and tolerability and to assess the efficacy of 100 mg, 200 mg, and 300 mg BID dextofisopam compared with placebo in female outpatients with diarrhea-predominant or alternating irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
This is a double-blind, randomized , placebo-controlled Phase 2b study of the safety, tolerability, and efficacy of 100, 200 and 300 mg BID dextofisopam in female patients suffering from diarrhea-predominant or alternating-Irritable Bowel Syndrome. (d-IBS or a-IBS.) Approximately 120 patients will be enrolled in each of the 4 arms of the study which will be conducted in up to 70 clinical sites in the USA. The patients will; be stratified by diagnosis.

Outpatient females, 18 to 65 years old will be enrolled in the study if diagnosed with d-IBS or a-IBS after having been screened during up to 17 days prior to enrollment (including colonoscopy if not done within the last 5 years) and found to have no organic disease that might have caused their complaints of abdominal pain or discomfort which when started was associated with a change in stool frequency or form and/or improves with defecation.

Patients will be instructed to take 3 capsules of the blinded study drug twice a day by mouth and to record by an interactive voice response system (IVRS ) any change in their symptoms. Patients who meet all the Inclusion and Exclusion criteria will be evaluated at baseline (one day prior to taking study drug ) including laboratory determinations including a pregnancy test for women of childbearing potential, vital signs, electrocardiogram ( ECG), recording of adverse events(AE's) and filling out the IBS Quality of Life Questionnaire( IBSQOL ), the Work Productivity and Activity Impairment Questionnaire-IBS Version ( WPAI:IBS )and the Hospital l Anxiety and Depression Questionnaire ( HAD).

Enrolled patients will have 12 weeks of double-blind treatment followed by a 28 day post treatment period.

Symptoms will be recorded daily

. Patients will visit the investigating site at weeks 4, 8 and 12 after the baseline visit and the procedures performed at baseline will be repeated A post treatment visit will occur 28 days after discontinuing study drug. Vital signs, AE's, concomitant medications and daily and weekly symptom assessment via IVRS will be recorded.

ELIGIBILITY:
Ages Eligible for Study: 18 Years - 65 Years, Genders Eligible for Study: Female

Inclusion Criteria:

* 1. Outpatient post-menopausal or no pregnant females,18 to 65 years old
* 2. Irritable bowel syndrome, which meet the Rome III criteria for IBS of the diarrhea-predominant or the alternating subtype
* 3. Able to give informed consent
* 4 Willingness to make daily calls on a touch-tone telephone

Exclusion Criteria:

* 1. Clinically significant abnormality on the screening tests.
* 2. Use of any other investigational drug within 30 days before screening visit.
* 3. Serious underlying diseases, including psychiatric disorders or current history of conditions affecting bowel habits
* 4. Previous treatment with tofisopam Related drugs.
* 5. History or presence of clinically significant medical disease that might compromise the study or be detrimental to the patient, such as
* 6. Subject has exclusively constipation-predominant IBS.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The percentage of weeks for which patients record adequate overall relief of IBS symptoms during the double blind period (12 weeks of treatment). | June 07 thru August 09

CONTACTS AND LOCATIONS:
Overall Officials: S Colin Neill, Study Chair — President and CFO, Pharmos
Locations (79):
- United States (79):
  - Alliance Clinical Research, Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Mobile Medical and Diagnostic Center, Mobile, Alabama
  - Radiant Research, Phoenix Southwest, Chandler, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Providence Clinical Research, Burbank, California
  - Discovery Clinical Research, Encinitas, California
  - Digestive and Liver Disease Specialists, Garden Grove, California
  - Community Clinical Trials, Orange, California
  - Advance Clinical Research Institute, Orange, California
  - Northern California Research, Sacramento, California
  - Medical Associates Research Group, San Diego, California
  - Westlake Medical Research, Westlake Village, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Rx Clinical Trials, Washington D.C., District of Columbia
  - Meridien Research, Brooksville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Genesis Research International, Longwood, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, LLC, Orlando, Florida
  - The Clinical Research Center of Northwest Florida, Panama City, Florida
  - ACCORD Clinical Research, LLC, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Perimeter Institute for Clinical Research, Inc. (PICR), Atlanta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Heartland Research Associates, LLC, Arkansas City, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Trover Health System, Madisonville, Kentucky
  - Clinical Trials of America, Shreveport, Louisiana
  - Maryland Digestive Disease Research, LLC, Laurel, Maryland
  - Capital Gastroenterology Consultants, PA, Silver Spring, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Gastrointestinal Associates, Jackson, Mississippi
  - Meridan Clinical Research, Omaha, Nebraska
  - Digestive Disease Specialists, Las Vegas, Nevada
  - New Mexico Clinical Research & Osteoporosis Center, Inc, Albuquerque, New Mexico
  - Long Island Clinical Research Associates, Great Neck, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Winthrop University Hospital, Mineola, New York
  - The Weill Medical College Of Cornell University, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Cumberland Research Associates, LLC., Fayetteville, North Carolina
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - Clinical Trials of America, Winston-Salem, North Carolina
  - Medical Frontiers, LLC, Carlisle, Ohio
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Digestive Health Network, Cincinnati, Ohio
  - Gastroenterology Research Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Gastrointestinal & Liver Diseases Consultants, PC, Dayton, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Aquilo Research, Yukon, Oklahoma
  - TriValley Primary Care-Pennridge, Perkasie, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - TriCities Medical Research, Bristol, Tennessee
  - ClinSearch, Chattanooga, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
  - Austin Gastroenterology, PA, Austin, Texas
  - Radiant Research of Dallas-North, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Sun Research Institute, San Antonio, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Gastroenterology Clinic of San Antonio, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Professional Place Medical Group, LLC, Chesapeake, Virginia
  - New River Valley Research Institute, Christiansburg, Virginia
  - National Clinical Recruiters, Inc, Richmond, Virginia
  - Wenatchee Valley Medical Center, Wenatchee, Washington